CLINICAL TRIAL: NCT01014208
Title: Ofatumumab Versus Rituximab Salvage Chemoimmunotherapy Followed by Autologous Stem Cell Transplant (ASCT) in Relapsed or Refractory Diffuse Large B Cell Lymphoma (DLBCL)
Brief Title: Ofatumumab Versus Rituximab Salvage Chemoimmunotherapy Followed by Autologous Stem Cell Transplant in Relapsed or Refractory Diffuse Large B Cell Lymphoma
Acronym: ORCHARRD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110928
Record Dates: First submitted 2009-11-04; First posted 2009-11-16 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-02

CONDITIONS: Lymphoma, Large-Cell, Diffuse
Keywords: The All Ireland Cooperative Oncology Research Group; GELTAMO; National Cancer Research Institute Lymphoma Clinical Studies Group; Genmab; ofatumumab; Japan Clinical Oncology Group; Oncology; Polish Lymphoma Research Group; Salvage chemotherapy; refractory; HOVON; DVD; relapsed; safety; efficacy; DHAP; rituximab; Autologous Stem Cell Transplant; Dutch-Belgian Cooperative Trial Group for Hematology-Oncology; Grupo Espanol de Linfomas; Nordic Lymphoma Group
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Neoplasms; Recurrence | interventions — ofatumumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OFATUMUMAB + DHAP CHEMOTHERAPY REGIMEN (Experimental): This study is a parallel arm study, with ofatumumab + DHAP. The Investigators are required to prospectively choose to treat all of their subjects with either DHAP chemotherapy regimens in combination with ofatumumab. All subjects will receive the same ofatumumab regimen and dose.
  Interventions: Drug: OFATUMUMAB + DHAP
- RITUXIMAB + DHAP CHEMOTHERAPY REGIMEN (Active Comparator): This study is a parallel arm study, with rituximab + DHAP. The Investigators are required to prospectively choose to treat all of their subjects with either DHAP chemotherapy regimens in combination with rituximab. All subjects will receive the same rituximab regimen and dose.
  Interventions: Drug: RITUXIMAB + DHAP

INTERVENTIONS:
Drug: OFATUMUMAB + DHAP — 3 cycles of treatment will be administered. Each cycle will last 21 days. ofatumumab dose: cycle 1, day 1 - 1000 mg; cycle 1, day 8 - 1000 mg; cycle 2, day 1 and cycle 3, day 1 - 1000 mg. DHAP regimen: dexamethasone - 40 mg on days 1, 2, 3, and 4 of dosing cycle; cisplatin - 100 mg/m2/24hrs continuous on day 1 of dosing cycle; cytarabine - 2g/m2 q12 hrs (2 doses) on day 2 of dosing cycle.
  Arms: OFATUMUMAB + DHAP CHEMOTHERAPY REGIMEN
Drug: RITUXIMAB + DHAP — 3 cycles of treatment will be administered. Each cycle will last 21 days. rituximab dose: cycle 1, day 1 - 375 mg/m2; cycle 1, day 8 - 375 mg/m2; cycle 2, day 1 and cycle 3, day 1 - 375 mg/m2. DHAP regimen: dexamethasone - 40 mg on days 1, 2, 3, and 4 of dosing cycle; cisplatin - 100 mg/m2/24hrs continuous on day 1 of dosing cycle; cytarabine - 2g/m2 q12 hrs (2 doses) on day 2 of dosing cycle.
  Arms: RITUXIMAB + DHAP CHEMOTHERAPY REGIMEN

SUMMARY:
This study is being conducted to compare the efficacy and safety of ofatumumab in addition to salvage chemotherapy versus rituximab in addition to salvage chemotherapy in CD20 positive DLBCL subjects relapsing, or with persistent disease, after first-line treatment with rituximab combined with an anthracycline-based chemotherapy regimen and be eligible for ASCT.

DETAILED DESCRIPTION:
As rituximab-based regimens have become standard first-line treatment in CD20 positive DLBCL, the efficacy of rituximab combined with salvage chemotherapy in the second-line setting has decreased and there is a need for new therapies in patients progressing or relapsing after first-line rituximab-based therapy. Replacement of rituximab with ofatumumab in the second-line setting, following progression/relapse after first-line rituximab-containing regimens, offers the potential to overcome relative or complete rituximab resistance and thus improve response rates, the ability to proceed to consolidative HDT/ASCT, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with CD20 positive DLBCL or grade 3b follicular lymphoma (FL) at original diagnosis.
* Refractory to, or relapsed following, first-line treatment with rituximab combined with anthracycline- or anthracenedione-based chemotherapy as defined by the protocol.
* CT with involvement of 2 or more clearly demarcated lesions/ nodes with a long axis > 1.5 cm and short axis >= 1.0cm or 1 clearly demarcated lesion/ node with a long axis > 2.0 cm and short axis >= 1.0 cm.
* Baseline FDG-PET scans must demonstrate positive lesions compatible with CT defined anatomical tumor sites.
* Age 18 yrs or older.
* ECOG performance status of 0, 1 or 2.
* Eligible for high dose chemotherapy and ASCT.
* Resolution of toxicities from first-line therapy to a grade that in the opinion of the investigator does not contraindicate study participation.
* Signed written informed consent.

Exclusion Criteria:

* Previous cancer therapy for lymphoma, with the exception of first-line rituximab/ anthracycline- or anthracenedione-based chemotherapy, monotherapy rituximab prior to or combined with first-line chemotherapy, as maintenance therapy, and radiotherapy in a limited field or as a part of the first-line treatment plan.
* Any anti-cancer therapy, except limited field radiotherapy, within 2 weeks prior to start of study therapy.
* Planned post-randomization chronic glucocorticoid use (limited acute use is allowed and defined by the protocol) unless administered as therapy for mild COPD or asthma.
* Clinically significant cardiac disease, active or chronic infections, serious significant diseases, other cancer within last 5 years. History of significant cerebrovascular disease.
* Prior treatment with anti-CD20 monoclonal antibodies with the exception of rituximab.
* Abnormal/ inadequate WBC count, liver, and kidney function.
* Pregnant or lactating women or female patients of child-bearing potential (or male patients with such partners) not willing to use adequate contraception during and up to 1 year following dosing completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2010-03; Primary Completion 2014-02 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (139):
- United States (15):
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Westwood, Kansas
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Chaple Hill, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Seattle, Washington
- Argentina (3):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
- Austria (5):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- Belgium (6):
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Yvoir
- China (10):
  - GSK Investigational Site, Fuzhou, Fujian
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Jianan, Shandong
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Jiang Su Province
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
- Czechia (2):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
- Denmark (2):
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Copenhagen
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (3):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Tampere
- Germany (4):
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, Athens, Greece
- Hungary (6):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Kaposvár
  - GSK Investigational Site, Szeged
  - GSK Investigational Site, Szombathely
- India (3):
  - GSK Investigational Site, Ludhiana
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Vellore
- Ireland (3):
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Galway
  - GSK Investigational Site, James Street
- Israel (2):
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
- Japan (16):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Akita
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokushima
  - GSK Investigational Site, Tokyo
- Netherlands (14):
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Hoofddorp
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Sittard-geleen
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Zwolle
- GSK Investigational Site, Oslo, Norway
- Poland (5):
  - GSK Investigational Site, Chorzów
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- GSK Investigational Site, Singapore, Singapore
- South Korea (2):
  - GSK Investigational Site, Jellanamdo
  - GSK Investigational Site, Seoul
- Spain (7):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Salamanca
- Sweden (4):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- GSK Investigational Site, Bangkok, Thailand
- United Kingdom (19):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Blackpool
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Cheltenham
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Headington, Oxford
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Northwood
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, Southampton
  - GSK Investigational Site, Whitchurch, Cardiff
  - GSK Investigational Site, Wolverhampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were refractory to, or had relapsed following, first-line treatment with rituximab in combination with an anthracycline- or anthracenedione-containing chemotherapy regimen, and who were eligible for autologous stem cell transplant (ASCT), were eligible for enrollment.
Pre-assignment Details: Eligible participants were randomized to receive either rituximab or ofatumumab in addition to salvage chemotherapy.
Groups:
- Rituximab + Chemotherapy: Participants received 3 cycles (21 days per cycle) of rituximab combined with salvage chemotherapy (SC): either the DHAP regimen (3 cycles of dexamethasone, cytarabine, cisplatin [DHAP]) or the DVD regimen (DHAP-VIM [etoposide, ifosfamide, mesna, methotrexate]-DHAP). Rituximab (375 milligrams per meters squared [mg/m^2]) was infused intravenously (IV) on Day (D) 1 (or up to 3 days prior to D1) and D8 (+/-2 days) of Cycle 1 of the SC, and then on D1 only of Cycles 2 and 3. The DHAP regimen (SC) contained: dexamethasone (40 mg/day) administered orally or IV on Days 1, 2, 3, or 4 of each cycle; cisplatin (100 mg/m^2/day) as an IV continuous infusion on D1 of each cycle; and cytarabine 2 grams (g)/m^2 over 3 hours every 12 hours (2 doses) for each infusion on D2 of each cycle. VIM: etoposide (90 mg/m^2 IV on Days 1, 3, and 5), ifosfamide (1200 mg/m^2 IV on Days 1, 2, 3, 4, and 5), mesna (10 or 20 mg/kilogram [kg] IV on Days 1, 2, 3, 4, and 5), methotrexate (30 mg/m^2 IV on Days 1 and 5).
- Ofatumumab + Chemotherapy: Participants received 3 cycles (21 days per cycle) of ofatumumab combined with SC: either the DHAP regimen (three cycles of DHAP) or the DVD regimen (DHAP-VIM-DHAP). Ofatumumab (1000 mg/1000 milliliter [mL]) was infused IV on Day 1 (or up to 3 days prior to Day 1) and Day 8 (+/-2 days) of Cycle 1 of the SC, and then on Day 1 only of Cycles 2 and 3. The DHAP regimen (SC) contained: dexamethasone (40 mg/day) administered orally or IV on Days 1, 2, 3, or 4 of each cycle; cisplatin (100 mg/[m^2]/day) as an IV continuous infusion on Day 1 of each cycle; and cytarabine 2 g/m^2 over 3 hours every 12 hours (2 doses) for each infusion on Day 2 of each cycle. VIM: etoposide (90 mg/m^2 IV on Days 1, 3, and 5), ifosfamide (1200 mg/m^2 IV on Days 1, 2, 3, 4, and 5), mesna (10 or 20 mg/kg IV on Days 1, 2, 3, 4, and 5), methotrexate (30 mg/m^2 IV on Days 1 and 5).
Period: Overall Study
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy
Started | 225 | 222
Intent-to-Treat Population | 223 | 222
Completed | 131 | 122
Not Completed | 94 | 100
Not completed — Lost to Follow-up | 2 | 5
Not completed — Participant Withdrew Consent | 12 | 12
Not completed — Did Not Receive Study Drug | 2 | 0
Not completed — Study Closed/terminated | 78 | 83

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy | Total
Number analyzed (Participants) | 223 | 222 | 445
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (12.22) | 55.2 (10.80) | 54.3 (11.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 85 | 173
  Male | 135 | 137 | 272
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 4 | 4 | 8
  American Indian or Alaska Native | 0 | 1 | 1
  Asian - Central/South Asian Heritage | 3 | 4 | 7
  Asian - East Asian Heritage | 24 | 31 | 55
  Asian - Japanese Heritage | 19 | 22 | 41
  Asian - South East Asian Heritage | 4 | 4 | 8
  Asian - Mixed Race | 0 | 1 | 1
  White - Arabic/North African Heritage | 1 | 1 | 2
  White - White/Caucasian/European Heritage | 168 | 151 | 319
  Missing | 0 | 3 | 3
Number of participants with the indicated SaaIPI scores [Number; unit: Participants] — The secondary age adjusted international prognostic index (SaaIPI) is assessed according to the absence or presence of 3 risk factors (RFs) at the start of Screening: Eastern Cooperative Oncology Group performance status greater than 1, lactate dehydrogenase level greater than the upper level of normal, and Ann Arbor stage II or IV disease. The presence of 0, 1, or more than 1 RFs corresponds to a SaaIPI score reflecting low, intermediate, and high risk of disease progression.
  Participants
    0 or 1 | 136 | 133 | 269
    2 or 3 | 87 | 89 | 176
Number of participants in the indicated categories per best response to first-line treatment [Number; unit: Participants] — Late relapsers are those participants with a complete response (CR: complete disappearance of all detectable clinical evidence of disease/disease-related symptoms) following first line treatment which lasts >12 months from diagnosis. Early relapsers/refractory are those participants with a CR <= 12 months, PR (>=50% decrease from Baseline in the sum of the product of the diameters of target lesions), SD (failure to attain CR or PR; no fulfillment of PD), or PD (disease that has grown or spread) after first-line treatment.
  Participants
    Late relapsers | 66 | 63 | 129
    Early relapsers/Refractory | 157 | 159 | 316

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival as Assessed by Independent Reviewers
Description: Progression-free survival is defined as the interval of time from the randomization date until the date of stable disease (SD; failure to attain the criteria needed for a CR or PR and no fulfillment of the criteria for progressive disease [PD]) after two cycles of salvage chemotherapy, progression, or death, whichever occurs first. Disease progression was based on the assessments of independent reviewers for the disease under study. Disease progression was based on imaging data via the Revised Response Criteria for Malignant Lymphoma (RRCML).
Time Frame: From randomization until the date of stable disease after two cycles of salvage chemotherapy, progression, or death (assessed for up to 5 years)
Population: Intent-to-Treat (ITT) Population: all participants who were randomized and commenced study therapy (at least one dose of a study drug)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy
Number analyzed (Participants) | 223 | 222
Months | 2.14 [1.64 to 4.37] | 1.81 [1.54 to 2.53]
Statistical Analysis 1: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Test type: Superiority or Other; p = 0.333, Stratified Log-rank test — p-value from stratified log-rank test are adjusted for stratification factors; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.89 to 1.42] — The Pike estimator was the statistical method used to estimate the hazard ratio

2. Secondary Outcome: Number of Participants With Overall Response (OR) and Complete Response (CR) After Salvage Chemoimmunotherapy
Description: OR is defined as the number of participants achieving either a complete response (CR) or a partial response (PR). CR is defined as the complete disappearance of all detectable clinical evidence of disease and disease-related symptoms. PR is defined as at least a 50% decrease from Baseline in the sum of the product of the diameters of target lesions. RRCML was used to assess CR and PR.
Time Frame: At completion of up to 3 cycles of salvage chemoimmunotherapy (assessed up to 9 weeks)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy
Number analyzed (Participants) | 223 | 222
Participants
  Independent reviewer-assessed OR | 94 | 84
  Independent reviewer-assessed CR | 48 | 34
Statistical Analysis 1: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Test type: Superiority or Other; p = 0.4053, Cochran-Mantel-Haenszel — p-value for the test of Odds Ratio being 1; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.56 to 1.24] — For Category title- Independent reviewer-assessed OR
Statistical Analysis 2: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Test type: Superiority or Other; p = 0.1167, Cochran-Mantel-Haenszel — p-value for the test of Odds Ratio being 1; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.39 to 1.10] — For Category title- Independent reviewer-assessed CR

3. Secondary Outcome: Number of Participants With Overall Response (OR) and Complete Response (CR) Three Months After Autologous Stem Cell Transplant
Description: as for outcome 2
Time Frame: At 3 months after completion of autologous stem cell transplantation (ASCT) (assessed up to 6 months)
Population: ITT Population. Only participants completing HDT/ASCT are included.
Measure: Number; unit: Participants
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy
Number analyzed (Participants) | 83 | 74
Participants
  Independent reviewer-assessed OR | 57 | 53
  Independent reviewer-assessed CR | 44 | 43
Statistical Analysis 1: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Test type: Superiority or Other; p = 0.8209, Cochran-Mantel-Haenszel — p-value for the test of Odds Ratio being 1; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.55 to 2.43] — For Category title- Independent reviewer-assessed OR
Statistical Analysis 2: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Test type: Superiority or Other; p = 0.6313, Cochran-Mantel-Haenszel — p-value for the test of Odds Ratio being 1; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.62 to 2.43] — For Category title- Independent reviewer-assessed CR

4. Secondary Outcome: Event-free Survival
Description: Event-free survival is defined as the time from randomization to progressive disease (PD; disease whose course is growth, or spread of the disease), stable disease (SD; failure to attain the criteria needed for a CR or PR and no fulfillment of the criteria for PD) after completion of 2 cycles of therapy, commencement of a new treatment for diffuse large B cell lymphoma (DLBCL) (e.g., radiotherapy), or death from any cause, whichever occurs first. Disease progression was based on the assessments of independent reviewers for the disease under study. Disease progression was based on imaging data via the Revised Response Criteria for Malignant Lymphoma (RRCML).
Time Frame: From randomization to progressive disease, stable disease after completion of 2 cycles of therapy, commencement of a new treatment for DLBCL, or death due to any cause (assessed for up to 5 years)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy
Number analyzed (Participants) | 223 | 222
Months | 1.84 [1.61 to 2.50] | 1.74 [1.54 to 2.23]
Statistical Analysis 1: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Test type: Superiority or Other; p = 0.346, Stratified log-rank test — p-value from stratified log-rank test are adjusted for stratification factors; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.90 to 1.36] — Confidence Interval estimated using the Brookmeyer-Crowley method. HR are estimated using Pike estimator. A hazard ratio <1 indicates a lower probability of recovery with Ofatumumab compared to Rituximab. HR was adjusted for stratification factors

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death due to any cause. Participants who were still alive by the end of the study were censored.
Time Frame: From randomization to death due to any cause (assessed for up to 5 years)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy
Number analyzed (Participants) | 223 | 222
Months | 13.17 [10.02 to 14.98] | 13.86 [10.91 to 22.41]
Statistical Analysis 1: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Test type: Superiority or Other; p = 0.377, Stratified log-rank test — p-value from stratified log-rank test are adjusted for stratification factors; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.70 to 1.15] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Number of Participants With the Ability to Mobilize at Least 2 Million Cluster of Differentiation (CD)34+ Cells Per Kilogram From Peripheral Blood
Description: Stem cell mobilization is the process of stimulating the hematopoietic stem cells (CD34+) to move out of the bone marrow and into the bloodstream, where they can be collected via a process called apheresis. Successful mobilization is defined as the collection of >2*10^6 CD34+ cells/kg. Only those participants, who commenced harvest, following the administration of rituximab or ofatumumab in combination with DHAP combination chemotherapy, were assessed. The number of participants with adequate harvest of CD34+ stem cells (at least 2*10^6 CD34+ cells/kg) after dosing of salvage therapy in Cycle 2 and Cycle 3 was analyzed.
Time Frame: During Cycles 2 and/or 3 (Weeks 4-9)
Population: ITT Population. Only participants commencing leukapheresis are included.
Measure: Number; unit: Participants
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy
Number analyzed (Participants) | 134 | 125
Participants | 121 | 120
Statistical Analysis 1: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Test type: Superiority or Other; p = 0.1161, Cochran-Mantel-Haenszel — p-value for the test of Odds Ratio being 1; Odds Ratio (OR) = 2.57, 95% CI 2-sided [0.83 to 9.50]

7. Secondary Outcome: Number of Participants Completing Autologous Stem Cell Transplant (ASCT)
Description: The number of participants who completed ASCT is reported.
Time Frame: Approximately 4 to 6 weeks following Cycle 3 (assessed up to 3 months)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy
Number analyzed (Participants) | 223 | 222
Participants | 83 | 74
Statistical Analysis 1: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Test type: Superiority or Other; p = 0.4481, Cochran-Mantel-Haenszel — p-value for the test of Odds Ratio being 1; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.56 to 1.27] — Statistics are presented for Completion rate

8. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-General (FACT-G) During Treatment
Description: The FACT-G was developed by the Functional Assessment of Chronic Illness Therapy (FACIT) group for use in adults in a wide range of oncology clinical trial populations. The 27 items of the FACT-G are scored in the following domains: Physical Well-being (7 items), Social/Family Wellbeing (7 items), Emotional Well-being (6 items), and Functional Well-being (7 items). Participants responded to the items on a five-point Likert scale ranging from 0, "Not at all" to 4, "Very much." The total score ranges from 0 to 108; higher scores indicate a better patient-reported outcome/quality of life. Participants were asked to think back over the past week when responding to the items.
Time Frame: Baseline and the end of the treatment period (until approximately 4 to 6 weeks following Cycle 3 [assessed up to 3 months])
Population: ITT Population. Only those participants who provided data were assessed.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy
Number analyzed (Participants) | 172 | 175
scores on a scale | -2.561 (0.7671) | -2.591 (0.7696)
Statistical Analysis 1: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Test type: Superiority or Other; p = 0.978, ANCOVA; Mean Difference (Final Values) = 0.030, 95% CI 2-sided [-2.110 to 2.170]

9. Secondary Outcome: Change From Baseline in the Functional Assessment of Cancer Therapy Lymphoma Trial Outcome Index (FACT-Lym TOI) Total Score During Treatment
Description: The FACT-Lym TOI is a measure that combines the FACT-Lym subscale (15 items; responses to each item range from 0, "Not at all" to 4, "Very much") with two domains taken from the FACT-G (responses to each item range from "Not at all " to "Very much"): Physical Well-being (7 items: lack of energy, nausea, meeting family needs, pain, side effects, feels ill, spends time in bed) and Functional Well-being (7 items: ability to work, work fulfilment, ability to enjoy life, illness acceptance, ability to sleep well, enjoying things done for fun, satisfaction with quality of life). This index is designed to be sensitive to changes in treatment regimens. The total FACT-Lym TOI score ranges from 0 to 116; higher scores indicate a better patient-reported outcome/quality of life. Participants were asked to think back over the past week when responding to the items.
Time Frame: as for outcome 8
Population: ITT Population. Only those participants who provided data were assessed.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy
Number analyzed (Participants) | 172 | 174
scores on a scale | -2.028 (0.9196) | -3.156 (0.9204)
Statistical Analysis 1: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Test type: Superiority or Other; p = 0.387, ANCOVA; Mean Difference (Final Values) = 1.129, 95% CI 2-sided [-1.434 to 3.691]

10. Secondary Outcome: Time to Neutrophil and Platelet Recovery After Each Cycle of Salvage Chemotherapy
Description: Neutrophil (absolute neutrophil count [ANC]) recovery is defined as ANC >=0.5*10^9/Liter and increasing, and platelet (PLT) recovery is defined as PLT >=10*10^9/Liter and increasing. For each cycle, time to ANC recovery is defined as the time from the first dose to the first ANC >=0.5*10^9/Liter and increasing after the nadir in the cycle. For each cycle, time to PLT recovery is defined as the time from the first dose to the first PLT >=10*10^9/L and increasing after the nadir in the cycle.
Time Frame: From the start of each cycle for a maximum of 5 weeks per cycle (assessed during treatment period of Baseline up to approximately 3 months)
Population: Safety Population. Only those participants available for analysis in the given cycle were assessed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy
Number analyzed (Participants) | 223 | 222
days
  Neutrophils, Cycle 1, n=223, 222 | 8.0 [6.0 to 13.0] | 11.0 [8.0 to 13.0]
  Neutrophils, Cycle 2, n=196, 199 | 8.0 [6.0 to 10.0] | 11.0 [9.0 to 13.0]
  Neutrophils, Cycle 3, n=137, 129 | 10.0 [6.0 to 12.0] | 7.0 [5.0 to 10.0]
  Platelets, Cycle 1, n=223, 222 | 13.0 [12.0 to 13.0] | 12.0 [12.0 to 13.0]
  Platelets, Cycle 2, n=196, 199 | 13.0 [12.0 to 13.0] | 13.0 [12.0 to 13.0]
  Platelets, Cycle 3, n=137, 129 | 13.0 [12.0 to 14.0] | 13.0 [12.0 to 14.0]
Statistical Analysis 1: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Statistics are presented for Category-Neutrophils, Cycle 1. Confidence Interval (CI) estimated using the Brookmeyer-Crowley method. HR are estimated using the Pike estimator. A hazard ratio <1 indicates a lower probability of recovery with Ofatumumab compared to Rituximab. HR was adjusted for stratification factors; Test type: Superiority or Other; p = 0.479, Stratified Log-Rank — p-value from stratified log-rank test are adjusted for stratification factors; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.74 to 1.16]
Statistical Analysis 2: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Statistics are presented for Category-Neutrophils, Cycle 2. Confidence Interval (CI) estimated using the Brookmeyer-Crowley method. HR are estimated using the Pike estimator. A hazard ratio <1 indicates a lower probability of recovery with Ofatumumab compared to Rituximab. HR was adjusted for stratification factors; Test type: Superiority or Other; p = 0.059, Stratified Log-Rank — p-value from stratified log-rank test are adjusted for stratification factors; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.64 to 1.02]
Statistical Analysis 3: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Statistics are presented for Category-Neutrophils, Cycle 3. Confidence Interval (CI) estimated using the Brookmeyer-Crowley method. HR are estimated using the Pike estimator. A hazard ratio <1 indicates a lower probability of recovery with Ofatumumab compared to Rituximab. HR was adjusted for stratification factors; Test type: Superiority or Other; p = 0.451, Stratified Log-Rank — p-value from stratified log-rank test are adjusted for stratification factors; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.83 to 1.48]
Statistical Analysis 4: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Statistics are presented for Category-Platelets, Cycle 1. Confidence Interval (CI) estimated using the Brookmeyer-Crowley method. HR are estimated using the Pike estimator. A hazard ratio <1 indicates a lower probability of recovery with Ofatumumab compared to Rituximab. HR was adjusted for stratification factors; Test type: Superiority or Other; p = 0.597, Stratified Log-Rank — p-value from stratified log-rank test are adjusted for stratification factors; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.86 to 1.29]
Statistical Analysis 5: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Statistics are presented for Category-Platelets, Cycle 2. Confidence Interval (CI) estimated using the Brookmeyer-Crowley method. HR are estimated using the Pike estimator. A hazard ratio <1 indicates a lower probability of recovery with Ofatumumab compared to Rituximab. HR was adjusted for stratification factors; Test type: Superiority or Other; p = 0.199, Stratified Log-Rank — p-value from stratified log-rank test are adjusted for stratification factors; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.70 to 1.10]
Statistical Analysis 6: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Statistics are presented for Category-Platelets, Cycle 3. Confidence Interval (CI) estimated using the Brookmeyer-Crowley method. HR are estimated using the Pike estimator. A hazard ratio <1 indicates a lower probability of recovery with Ofatumumab compared to Rituximab. HR was adjusted for stratification factors; Test type: Superiority or Other; p = 0.102, Stratified Log-Rank — p-value from stratified log-rank test are adjusted for stratification factors; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.93 to 1.59]

11. Secondary Outcome: Time to Engraftment After High-dose Therapy (HDT)/ASCT
Description: Engraftment is defined as 1) three consecutive days when the ANC is ≥0.5x109/L and 2) an unsupported platelet count of ≥20x109/L, and the engraftment date is the date that this occurs. If engraftment was not achieved by Day 42 or the last observation, engraftment was deemed to be a failure, and censoring took place at Day 42 or at the last observation.
Time Frame: From ASCT up to 42 days post-ASCT (Baseline up to approximately 4.5 months)
Population: Safety population. Only participants completing HDT/ASCT are included.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy
Number analyzed (Participants) | 83 | 74
Days | 24.0 [16.0 to NA] — The upper limit of the confidence interval cannot be calculated because there were too few events of engraftment. | NA [26.0 to NA] — The median cannot be calculated because there were too few events of engraftment The upper limit of the confidence interval cannot be calculated because there were too few events of engraftment.
Statistical Analysis 1: Comparison: Rituximab + Chemotherapy vs Ofatumumab + Chemotherapy; Test type: Superiority or Other; p = 0.035, Stratified Log-Rank — p-value from stratified log-rank test are adjusted for stratification factors; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.36 to 1.00] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected up to 60 days after the last dose of study treatment, or the commencement of high-dose chemotherapy, or anti-cancer therapy, whichever occurred first (up to approximately 16 study weeks).
Description: Serious adverse events (SAEs) and non-serious AEs were collected in members of the Safety Population, comprised of all participants who received at least one dose of study drug.
Arm/Group | Rituximab + Chemotherapy | Ofatumumab + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 115/223 | 118/222
Other Adverse Events (participants affected / at risk) | 217/223 | 215/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Chemotherapy (N=223) | Ofatumumab + Chemotherapy (N=222)
Febrile neutropenia (Blood and lymphatic system disorders) | 30 | 28
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 12
Neutropenia (Blood and lymphatic system disorders) | 7 | 6
Pancytopenia (Blood and lymphatic system disorders) | 1 | 5
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Sepsis (Infections and infestations) | 9 | 4
Neutropenic sepsis (Infections and infestations) | 4 | 8
Pneumonia (Infections and infestations) | 2 | 4
Device related infection (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 4 | 2
Infection (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 1 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 2
Pulmonary mycosis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 2 | 0
Abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Fungal endocarditis (Infections and infestations) | 1 | 0
Gastrointestinal candidiasis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Post procedural sepsis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 13 | 10
Nausea (Gastrointestinal disorders) | 9 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 5
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Ileal stenosis (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 12 | 11
Renal failure (Renal and urinary disorders) | 3 | 6
Renal impairment (Renal and urinary disorders) | 5 | 2
Renal injury (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Pyrexia (General disorders) | 11 | 8
Mucosal inflammation (General disorders) | 2 | 3
Fatigue (General disorders) | 0 | 3
General physical health deterioration (General disorders) | 1 | 2
Chest pain (General disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Blood creatinine increased (Investigations) | 5 | 12
Platelet count decreased (Investigations) | 2 | 7
Neutrophil count decreased (Investigations) | 1 | 3
Alanine aminotransferase increased (Investigations) | 0 | 2
White blood cell count decreased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0
Electrocardiogram change (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 4
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 6
Encephalopathy (Nervous system disorders) | 1 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 2
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 2
Thrombosis (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Ischaemia (Vascular disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Blindness (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Eyelid function disorder (Eye disorders) | 0 | 1
Ocular hypertension (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2
Completed suicide (Psychiatric disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Euthanasia (General disorders) | 0 | 1
Brachial plexopathy (Nervous system disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Secondary immunodeficiency (Immune system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Chemotherapy (N=223) | Ofatumumab + Chemotherapy (N=222)
Nausea (Gastrointestinal disorders) | 136 | 129
Vomiting (Gastrointestinal disorders) | 81 | 68
Constipation (Gastrointestinal disorders) | 65 | 76
Diarrhoea (Gastrointestinal disorders) | 70 | 50
Dyspepsia (Gastrointestinal disorders) | 24 | 16
Abdominal pain (Gastrointestinal disorders) | 19 | 17
Abdominal pain upper (Gastrointestinal disorders) | 14 | 12
Stomatitis (Gastrointestinal disorders) | 11 | 12
Anaemia (Blood and lymphatic system disorders) | 136 | 125
Thrombocytopenia (Blood and lymphatic system disorders) | 109 | 103
Neutropenia (Blood and lymphatic system disorders) | 71 | 67
Leukopenia (Blood and lymphatic system disorders) | 25 | 24
Febrile neutropenia (Blood and lymphatic system disorders) | 24 | 21
Fatigue (General disorders) | 80 | 74
Pyrexia (General disorders) | 69 | 60
Oedema peripheral (General disorders) | 30 | 31
Oedema (General disorders) | 21 | 24
Mucosal inflammation (General disorders) | 28 | 11
Chills (General disorders) | 24 | 13
Malaise (General disorders) | 17 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 57 | 58
Hypomagnesaemia (Metabolism and nutrition disorders) | 46 | 51
Hypocalcaemia (Metabolism and nutrition disorders) | 37 | 30
Hyponatraemia (Metabolism and nutrition disorders) | 25 | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 16 | 14
Hypophosphataemia (Metabolism and nutrition disorders) | 16 | 12
Platelet count decreased (Investigations) | 63 | 64
Blood creatinine increased (Investigations) | 31 | 45
White blood cell count decreased (Investigations) | 25 | 33
Neutrophil count decreased (Investigations) | 21 | 34
Weight increased (Investigations) | 22 | 22
Haemoglobin decreased (Investigations) | 18 | 21
Aspartate aminotransferase increased (Investigations) | 20 | 17
Alanine aminotransferase increased (Investigations) | 19 | 15
Weight decreased (Investigations) | 11 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 27
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 | 17
Hiccups (Respiratory, thoracic and mediastinal disorders) | 20 | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 12
Headache (Nervous system disorders) | 45 | 46
Dizziness (Nervous system disorders) | 31 | 23
Dysgeusia (Nervous system disorders) | 19 | 16
Rash (Skin and subcutaneous tissue disorders) | 19 | 48
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 34
Bone pain (Musculoskeletal and connective tissue disorders) | 14 | 12
Hypertension (Vascular disorders) | 14 | 18
Hypotension (Vascular disorders) | 11 | 20
Insomnia (Psychiatric disorders) | 24 | 28
Tinnitus (Ear and labyrinth disorders) | 21 | 14
Lethargy (Nervous system disorders) | 12 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 16
Flushing (Vascular disorders) | 7 | 12
Renal failure acute (Renal and urinary disorders) | 13 | 8
Renal impairment (Renal and urinary disorders) | 12 | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 13
Decreased appetite (Metabolism and nutrition disorders) | 54 | 56
Blood potassium decreased (Investigations) | 8 | 13
Blood lactate dehydrogenase increased (Investigations) | 12 | 8
Gamma-glutamyltransferase increased (Investigations) | 10 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.